#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | | Reporting and Analysis Plan for a single centre, single dose, open-label, randomised, 2-way crossover study in healthy Japanese male subjects to evaluate bioequivalence of daprodustat tablets (2 mg tablet vs. 4 mg tablet) (Part 1) and the food effect on the pharmacokinetics of daprodustat (Part 2) |
| <b>Compound Number</b> | : | GSK1278863 |
| <b>Effective Date</b> | : | 10-JUL-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207727.
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## RAP Author(s):

| Approver | Date | Approval Method |
|------------------------------------------------|------|-----------------|
| PPD | | |
| Biostatistics Group 2, Biomedical Data Science | s NA | NA |
| Japan | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Lead Programmer; Statistical Programming & Reporting Group, Biomedical Data Sciences Japan | 09-JUL-2018 | Pharma TMF |
| PPD | 00 1111 2010 | Dhama TME |
| Clinical Lead; Clinical Pharmacology Office | 09-JUL-2018 | Pharma TMF |
| PPD | 09-JUL-2018 | Pharma TMF |
| Clinical Scientist; Clinical Pharmacology Office | 0) JOE 2010 | Thaima Tivii |
| Operational Lead; Clinical Pharmacology Office | 09-JUL-2018 | Pharma TMF |
| Data Quality Lead; Data Practice Group,<br>Biomedical Data Sciences Japan | 09-JUL-2018 | Pharma TMF |
| PK Analyst; Clinical Pharmacology Office | 09-JUL-2018 | Pharma TMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Lead Authors Line Manager; Biostatistics Group 2, Biomedical Data Sciences Japan | 10-JUL-2018 | Pharma TMF |
| Lead Programmers Line Manager; Statistical Programming & Reporting Group, Biomedical Data Sciences Japan | 10-JUL-2018 | Pharma TMF |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | DN | 5 |
| 2. | SHIM | MARY OF | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | Objective(s) and Endpoint(s) | |
| | 2.2. | | Design | |
| | 2.3.<br>2.4. | Statistic | cal Hypotheses / Statistical Analyses | 9 |
| 3. | | | ALYSES | |
| | 3.1. | | Analyses | |
| | 3.2. | Final Ar | nalyses | 10 |
| 4. | ANAL | YSIS PO | PULATIONS | 11 |
| | 4.1. | | l Deviations | |
| 5. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | _ | S | |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | |
| | 5.3. | | ation of Covariates, Other Strata and Subgroups | 13 |
| | | 5.3.1. | Covariates and Other Strata | 13 |
| | 5.4. | Other C | Considerations for Data Analyses and Data Handling tions | 12 |
| | | Conven | lil0115 | 13 |
| 6. | STUE | Y POPU | LATION ANALYSES | 14 |
| | 6.1. | Overvie | w of Planned Study Population Analyses | 14 |
| | | 6.1.1. | | |
| 7. | SAFE | ΤΥ ΔΝΔΙ | YSES | 16 |
| ٠. | 7.1. | | Events Analyses | |
| | 7.1. | 7.1.1. | Details of Planned Adverse Events Summaries | |
| | 7.2. | | Laboratory Analyses | |
| | 1.2. | 7.2.1. | | |
| | 7.3. | | afety Analyses | |
| | 1.5. | 7.3.1. | | |
| | | 7.3.1. | Details of Flatified Other Safety Displays | 19 |
| 8. | | | NETIC ANALYSES | |
| | 8.1. | | cokinetic Analyses | |
| | | 8.1.1. | Endpoint / Variables | |
| | | | 8.1.1.1. Drug Concentration Measures | 20 |
| | | | 8.1.1.2. Derived Pharmacokinetic Parameters | <mark>20</mark> |
| | | 8.1.2. | Summary Measure | <mark>21</mark> |
| | | 8.1.3. | Population of Interest | <mark>21</mark> |
| | | 8.1.4. | Strategy for Intercurrent (Post-Randomization) Events | 21 |
| | | 8.1.5. | Statistical Analyses / Methods | |
| | | | 8.1.5.1. Statistical Methodology Specification | |
| | | 8.1.6. | Details of Planned Pharmacokinetic Displays | |

| 9. | REFE | RENCES | 25 |
|---|---|---|---|
| 10 | APPFI | NDICES | 26 |
| 10. | 10.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | 20 |
| | 10.1. | Protocol Population | 26 |
| | 10.2. | Appendix 2: Schedule of Activities | |
| | 10.2. | 10.2.1. Protocol Defined Schedule of Events | |
| | 10.3. | Appendix 3: Study Phases and Treatment Emergent Adverse | |
| | . 0.0. | Events | 28 |
| | | 10.3.1. Study Phases | |
| | | 10.3.1.1. Study Phases for Adverse Events | |
| | | 10.3.1.2. Study Phases for Concomitant Medication | |
| | 10.4. | Appendix 4: Data Display Standards & Handling Conventions | |
| | | 10.4.1. Reporting Process | |
| | | 10.4.2. Reporting Standards | |
| | | 10.4.3. Reporting Standards for Pharmacokinetic | |
| | 10.5. | Appendix 5: Derived and Transformed Data | 32 |
| | | 10.5.1. General | 32 |
| | | 10.5.2. Study Population | 32 |
| | | 10.5.3. Safety | |
| | 10.6. | Appendix 6: Reporting Standards for Missing Data | 34 |
| | | 10.6.1. Premature Withdrawals | |
| | | 10.6.2. Handling of Missing Data | 34 |
| | | 10.6.2.1. Handling of Missing and Partial Dates and | |
| | | Times | |
| | 10.7. | Appendix 7: Values of Potential Clinical Importance | |
| | | 10.7.1. Laboratory Values | |
| | | 10.7.2. ECG | |
| | 40.0 | 10.7.3. Vital Signs | 37 |
| | 10.8. | Appendix 8: Abbreviations & Trade Marks | |
| | | 10.8.1. Abbreviations | |
| | 40.0 | 10.8.2. Trademarks | |
| | 10.9. | Appendix 9: List of Data Displays | |
| | | 10.9.1. Data Display Numbering | |
| | | 10.9.2. Mock Example Shell Referencing | |
| | | 10.9.4. Study Population Tables | |
| | | 10.9.5. Safety Tables | |
| | | 10.9.6. Pharmacokinetic Tables | 42<br>45 |
| | | 10.9.7. Pharmacokinetic Figures | |
| | | 10.9.8. ICH Listings | |
| | 10 10 | Appendix 10: Example Mock Shells for Data Displays | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol GlaxoSmithKline Document Number 2017N354137\_00.

# **REVISION HISTORY**

Note that minor wording changes are not included in below.

| Reporting and Analysis Plan_207727_Amendment_Final_V1.1 [10-JUL-2018] | | | |
|---|---|---|---|
| Section # and Name | Description of Change | Brief Rationale | |
| 6.1 - Overview of<br>Planned Study<br>Population<br>Analyses | Listing of reasons for treatment discontinuation was added. | | eCRF screen was changed to capture treatment discontinuation. |
| 6.1.1- Details of<br>Planned Study<br>Population<br>Summaries | Removed the detail of summary display for race and racial combinations | | Corrections |
| 10.9 - Appendix 9:<br>List of Data<br>Displays | Table 1.5, Table 1.6 Listing 4, Listing 5 discontinuation added | Programming notes corrected. Listing for treatment | Corrections |
| | Listing 8, Listing 9 | IDSL/Example shell corrected | |
| | Table 3.7, Table 3.8 modified | Order of PK parameters in a title | |
| | Figure 3.9, Figure 3.10 modified | Order of PK parameters in a title | |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol (Dated: 12/Mar/2018) are outlined below. The change was intended to create some displays required by EudraCT with the "Enrolled" population.

| Protocol | |
|---|---|
| Section 9.3 Population for Analyses | |
| Population | Description |
| Enrolled | All subjects who signed the ICF |
| Safety | This population will be defined for each Part. |
| | · All randomised subjects who received at least one dose of study intervention. |
| PK | This population will be defined for each Part. |
| | · All subjects in the Safety population who had at least 1 non-missing PK |
| | assessment (Non-quantifiable [NQ] values will be considered as non-missing |
| | values). |
| | ' Di |
| Reporting & Analys | |
| Section 4. Ar | nalysis Populations |
| Population | Description |
| Screened | All subjects who signed the ICF |
| Enrolled | · All subjects who passed screening and entered the study. |
| | · Note screening failures (who never passed screening even if rescreened) and |
| | subjects screened but never enrolled into the study (Reserve, Not Used) are |
| | excluded from the Enrolled population as they did not enter the study. |
| Safety This population will be defined for each Part. | |
| · All randomised subjects who received at least one dose of study interve | |
| PK | This population will be defined for each Part. |
| | · All subjects in the Safety population who had at least 1 non-missing PK |
| | assessment (Non-quantifiable [NQ] values will be considered as non-missing |
| | values). |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Part 1 To determine the bioequivalence of daprodustat 2 mg tablet vs. 4 mg tablet in healthy Japanese male subjects. Part 2 To investigate the food effect on PK of daprodustat following a single dose of daprodustat in the fed and fasted | <ul> <li>Part 1 and 2</li> <li>Plasma PK parameters for daprodustat: AUC(0-t), Cmax, and the other parameters [AUC(0-inf), Tmax, t1/2, %AUCex, CL/F, Vz/F, kel and MRT]</li> </ul> |
| state in healthy Japanese male subjects. | |
| Secondary Objectives | Secondary Endpoints |
| Part 1 and 2 | Part 1 and 2 |
| To assess the safety and tolerability of<br>single dose of daprodustat following<br>administration of daprodustat in<br>healthy Japanese male subjects. | <ul> <li>Safety: Adverse events (AEs), clinical laboratory tests,<br/>vital signs (blood pressure, pulse and body temperature),<br/>and 12-lead electrocardiogram (ECG) parameters.</li> </ul> |

# 2.3. Study Design

| Overview of St | udy Design and Key F | eatures | |
|---|---|---|---|
| Design<br>Features | <ul> <li>This study consists of two parts; Part 1 is a single centre, single dose, open-label, randomised, 2-way crossover study in healthy Japanese male subjects. Part 2 is a single centre, single dose in the fed and fasted state, open-label, randomised, 2-way crossover study in healthy Japanese male subjects.</li> <li>In both part (Part 1 and Part 2), healthy subjects will have a screening visit within 30 days prior to the first dose of study treatment, two treatment periods, and re-visit 7 (±1) days after the second dose for follow-up. All subjects will be administered daprodustat as a single oral dose, with assessments conducted for up to 24 hours post-dose. Subjects will be housed in the Clinical Research Unit from Day -1 through Day 2 of each period. At least 5-day wash-out period will occur between each treatment period.</li> </ul> | | |
| Dosing | | vided into the study of Part 1 and<br>rt 1: A or B, Part 2: C or D) in the | d 2, and will be randomized to one efollowing table; |
| | <ul> <li>Part 1 (Bioequivalence part)</li> <li>Daprodustat 2 mg tablet x 2, single dose, in the fasted state</li> <li>Daprodustat 4 mg tablet x 1, single dose, in the fasted state</li> </ul> | | |
| | Group n | Period 1 | Period 2 |
| | A 26 | 2 mg tablet x 2 | 4 mg tablet x 1 |
| | B 26 4 mg tablet x 1 2 mg tablet x 2 | | |
| | • | a <b>rt)</b><br>4 mg tablet, single dose, in the fe<br>4 mg tablet, single dose, in the fa | |
| | Group n | Period 1 | Period 2 |
| | C 6 | 4 mg tablet x 1 (fed) | 4 mg tablet x 1 (fasted) |
| | D 6 | 4 mg tablet x 1 (fasted) | 4 mg tablet x 1 (fed) |
| | Blood sampling for PK analysis will be performed prior to dosing and until 24 hours post-<br>dose following each dose. The duration of each subject's participation will be<br>approximately 6 weeks from screening to the follow-up. | | |
| Time & Events | Refer to Appendix | 2: Schedule of Activities | |
| Treatment<br>Assignment | <ul> <li>Subjects will be assigned to one of two groups in accordance with the randomisation<br/>schedule generated by the Biomedical Data Sciences Department at GSK, prior to the<br/>start of the study, using validated internal software.</li> </ul> | | |
| Interim<br>Analysis | No interim analysis | s is planned. | |

## 2.4. Statistical Hypotheses / Statistical Analyses

#### Part 1:

The bioequivalence between daprodustat 2 mg tablet and 4 mg tablet will be demonstrated using a framework of statistical hypothesis testing. The ratio of the geometric means ( $\mu_{2mg}/\mu_{4mg}$ ) for AUC(0-t) and Cmax is the measure in the following statistical hypotheses:

 $H_0$  (null hypothesis) :  $\mu_{2mg}/\mu_{4mg} \le 0.80$  or  $\mu_{2mg}/\mu_{4mg} \ge 1.25$ 

 $H_1$  (alternative hypothesis) :  $0.80 < \mu_{2mg}/\mu_{4mg} < 1.25$ 

A judgment by 90% CI will be conducted in this study. The null hypothesis is rejected if the 90% confidence interval (CI) of  $\mu_{2mg}/\mu_{4mg}$  falls within a range of 0.80 to 1.25, which results a conclusion of the bioequivalence. This is equivalent to carrying out two one-sided tests of hypothesis at the 5% level of significance.

If the 90% CI of  $\mu_{2mg}/\mu_{4mg}$  doesn't fall within a range of 0.80 to 1.25 (i.e., null hypothesis is not rejected), the bioequivalence is established if the point estimate ( $\mu_{2mg}/\mu_{4mg}$ ) falls within a range of 0.90 to 1.11.

#### Part 2:

No formal statistical hypothesis will be tested.

# 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analysis is planned.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed the ICF. | Study Population |
| Enrolled | All participants who passed screening and entered the study. Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | |
| Safety | This population will be defined for each Part. All randomised participants who received at least one dose of study treatment. | Study Population,<br>Safety |
| Pharmacokinetic<br>(PK) | This population will be defined for each Part. All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). | PK |

Refer to Section 10.9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code Description | | Description | Order in TLF |
| | Part 1 (Schedule 1) | | |
| D1 | 2 mg x 2 | 2 mg x 2 | 1 |
| D2 | 4 mg x 1 | 4 mg x 1 | 2 |
| | Part 2 (Schedule 2) | | |
| D3 | 4 mg fed | 4 mg fed | 1 |
| D4 | 4 mg fasted | 4 mg fasted | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1.  $2mg \times 2 / 4mg \times 1$
- 2. fed / fasted

## 5.2. Baseline Definitions

Baseline definitions defined in the table are applicable to each period.

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asses | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | Screening Day -1 Day 1 (Pre-Dose) | | |
| Safety | | | | |
| Haematology | X | Χ | | Day -1 |
| Chemistry | X | Χ | | Day -1 |
| 12-lead ECG & Vital<br>Signs | Х | | Х | Day 1 (Pre-dose) |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries and statistical analyses. Additional covariates of clinical interest may also be considered.

| Category | Details |
|---|---|
| Covariates | See Section 8.1.5.1, describing pharmacokinetic analyses using statistical model |

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Schedule of Activities |
| 10.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition for the Subject Conclusion Record | Υ | | Υ |
| Treatment Status and Reasons for Discontinuation of Study Treatment | | | Υ |
| Screening Status and Reasons for Screen Failure | Y | | Υ |
| Number of Subjects Enrolled by Country and Site ID | Y | | |
| Planned and Actual Treatments | | | Υ |
| Protocol Deviations | · | | |
| Important Protocol Deviations | Y | | Υ |
| Inclusion/Exclusion Criteria Deviations | | | Υ |
| Population Analysed | | | |
| Subjects Excluded from PK Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Race and Racial Combinations | | | Υ |
| Age Ranges | Y | | |
| Medical Conditions and Concomitant Medications | | | |
| Medical Conditions | | | Υ |
| Concomitant Medications | | | Υ |
| Exposure | | | |
| Exposure to Study Treatment | | | Υ |
| Meal | | | |
| Meal start and end days/times on fed treatment | | | Υ |

#### NOTES:

• Y = Yes display generated.

## 6.1.1. Details of Planned Study Population Summaries

Summaries will be provided by Part (2 mg x 2 and 4 mg x 1 in Part 1, fed and fasted in Part 2), unless otherwise specified.

#### **Subject Disposition**

## Subject Disposition for the Subject Conclusion Record

The number and percentage of subjects who completed the study as well as subjects who withdrew from the study will be summarized. Reason for withdrawal will also be summarized for subjects who withdrew from the study. Only the total column will appear.

#### Screening Status and Reasons for Screen Failure

This will be based on Screened population. The number and percentage of subjects who passed screening and who failed screening and therefore were not entered into the study will be summarized along with the reasons for failure will be summarized for those subjects who failed screening. Only the total column will appear.

## Number of Subjects Enrolled by Country and Site ID

This will be based on Enrolled population. The number of subjects summarized by Country, Site ID and Investigator name will be presented. Only the total column will appear.

#### **Protocol Deviations**

#### Important Protocol Deviations

The number and percentage of subjects who had important protocol deviations defined as part of the protocol deviation management plan for the study, will be summarized. Only the total column will appear.

#### **Demographic and Baseline Characteristics**

#### Demographic Characteristics

The number and percentage of subjects or summary statistics will be provided for each demographic characteristic and only the total column will appear: Sex, Age (years), Age Group (years), Ethnicity, Race detail, Height, Weight, and Body Mass Index. Age Group (years) will be categorized into three ('≤18', '19-64', '≥65'). Each demographic characteristic will be summarized using the minimum set of summary statistics.

#### Age Ranges

This will be based on Enrolled population. The number and percentage of subjects within each age range category will be provided. Only the total column will appear. Only age ranges that are applicable to the study will be included (i.e., only '18-64 years'). This is based on the standard of EMA clinical trial results disclosure requirements.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

| Display Type | | Absolute | |
|---|---|---|---|
| | Sum | Individual | |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Y | | Y |
| All AEs by Maximum Intensity | Y | | |
| Drug-Related AEs by SOC and PT | Y | | |
| Drug-Related AEs by Maximum Intensity | Y | | |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Y |
| Serious and Other Significant AEs | | | |
| Serious AEs | | | Y |
| AEs Leading to Withdrawal from Study | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.1. Details of Planned Adverse Events Summaries

Summaries will be provided by Part (2 mg x 2 and 4 mg x 1 in Part 1, fed and fasted in Part 2), unless otherwise specified.

#### **Adverse Events (AEs)**

#### All AEs by SOC and PT

The number and percentage of subjects with all relevant adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### All AEs by Maximum Intensity by SOC and PT

The number and percentage of subjects with adverse events by intensity (e.g., mild, moderate, severe) will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

## Drug-related AEs by SOC and PT

The number and percentage of subjects with all drug-related adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Drug-related AEs by Maximum Intensity by SOC and PT

The number and percentage of subjects with drug-related adverse events by intensity (e.g., mild, moderate, severe) will be summarized by MedDRA System Organ Class and Preferred Term by treatment group and total. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

| Display Type | Absolute | | |
|---|---|---|---|
| | Sum | mary | Individual |
| | Т | F | L |
| Chemistry | | | |
| Chemistry Changes from Baseline | Υ | | |
| Chemistry Values | Y | | Υ |
| Chemistry Data Shifts from Baseline Relative to Normal Range | Υ | | |
| All Chemistry Data for Subjects with any Value of PCI | | | Υ |
| Chemistry Values of PCI | | | Υ |
| Haematology | | | |
| Haematology Changes from Baseline | Y | | |
| Haematology Values | Y | | Υ |
| Haematology Data Shifts from Baseline Relative to Normal Range | Υ | | |
| All Haematology Data for Subjects with any Value of PCI | | | Υ |
| Haematology Values of PCI | | | Υ |
| Urinalysis | | | |
| Urinalysis Concentration Changes from Baseline (Gravity and pH) | Υ | | |
| Urinalysis Data (Gravity and pH) | Υ | | Υ |
| Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) | Υ | | Y |
| Hepatobiliary (Liver) | | | |
| Liver Monitoring/Stopping Event Reporting | | | Υ |
| Medical Conditions for Subjects with Liver Stopping Events | | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.2.1. Details of Planned Clinical Laboratory Displays

Summaries will be provided by Part (2 mg x 2 and 4 mg x 1 in Part 1, fed and fasted in Part 2), unless otherwise specified.

#### Chemistry/Haematology Laboratory Tests

#### Laboratory Changes from Baseline and Values

Each quantitative laboratory test and the changes in value from baseline will be summarized at every assessed time point using n, mean, standard deviation, median, minimum, and maximum by treatment group.

#### Laboratory Data Shifts from Baseline Relative to Normal Range

The number and percentage of subjects with laboratory results within each normal range (Low, Normal, High) during each period will be summarized relative to their baseline category by laboratory test. The percentages are based on the number of subjects in the treatment group with data for the laboratory test at the specified planned time (n). Subjects are only counted once in the total column.

#### **Urinalysis Laboratory Tests**

#### *Urinalysis Concentration Changes from Baseline (Gravity and pH)*

Gravity and pH test and the changes in value from baseline will be summarized at every assessed time point using n, mean, standard deviation, median, minimum, and maximum by treatment group.

#### *Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen)*

The number and percentage of subjects with the above urinalysis results (character results) will be summarized by treatment group.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays.

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Υ | | | |
| ECG Values | Υ | | Y | Υ | | |
| All ECG Values for Subjects with any Value of PCI | | | Y | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | |
| All Vital Signs for Subjects with any Value of PCI | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.3.1. Details of Planned Other Safety Displays

Summaries will be provided by Part (2mg tablet x 2 and 4mg tablet x 1 in Part 1, fed state and fasted state in Part 2), unless otherwise specified.

#### **ECG**

#### ECG Findings

The number and percentage of subjects with ECG findings (ECG interpretation) will be summarized by treatment group.

#### ECG Values

Each ECG parameter value and the change from baseline will be summarized by treatment group at every assessed time point using n, mean, standard deviation, median, minimum, and maximum.

#### Vital Signs

#### Vital Signs

Each vital sign parameter and the changes in value from baseline will be summarized by treatment group at every assessed time point using n, mean, standard deviation, median, minimum, and maximum.

## 8. PHARMACOKINETIC ANALYSES

## 8.1. Pharmacokinetic Analyses

#### 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters of daprodustat will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t)<br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| AUC(0-inf)<br>(h*ng/mL) | The area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: AUC(0-inf) = AUC(0-t) + Ct / kel |
| Cmax<br>(ng/mL) | Maximum observed plasma concentration following each dose will be obtained directly from the concentration-time data. |
| Tmax (h) | The time to maximum observed plasma drug concentration following each dose will be obtained directly from the concentration-time data. |
| t1/2 (h) | Terminal half-life will be calculated as follows:<br>t1/2 = ln2 / kel |
| %AUCex (%) | The percentage of AUC(0-inf) obtained by extrapolation (%AUCex) will be calculated as follows: %AUCex = (AUC(0-inf) – AUC(0-t)) / AUC(0-inf) x 100 |
| CL/F<br>(mL/h) | Apparent clearance following oral dosing will be calculated as follows: CL/F = Dose / AUC(0-inf) |
| Vz/F<br>(mL) | Apparent volume of distribution after oral administration will be calculated as follows: Vz/F = Dose / (kel x AUC(0-inf)) |
| MRT<br>(h) | Mean residence time will be calculated as follows: MRT = AUMC(0-inf) / AUC(0-inf) |
| Tlast (h) | The time of the last measurable (positive) concentration. |
| kel | The first order rate constant associated with the terminal (log-linear) portion of the curve. |

| Parameter | Parameter Description |
|---|---|
| (lambda_z)<br>(/h) | |
| lambda_z_lo<br>wer | The lower limit on time for values to be included in the calculation of kel. |
| lambda_z_u<br>pper | The upper limit on time for values to be included in the calculation of kel. |
| #pts | The number of time points used in computing kel. |
| R-square | The goodness of fit statistic for the terminal elimination phase. |

#### NOTES:

- Additional parameters may be included as required.
- Kel is the terminal phase rate constant.
- Ct is the last observed quantifiable concentration.

## 8.1.2. Summary Measure

In Part 1, the ratio of geometric mean for AUC(0-t) and Cmax between daprodustat 2 mg tablet x 2 and 4 mg tablet x 1 will be used for the comparison between daprodustat 2mg tablet x 2 vs. daprodustat 4mg tablet x 1.

In Part 2, the ratio of geometric mean for AUC(0-t) and Cmax between fed and fasted state will be used for the comparison between the fed state vs. the fasted state.

## 8.1.3. Population of Interest

The pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

## 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events which may affect the evaluation of bioequivalence and food effect will not be anticipated.

#### 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Section 8.1.6: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

Derived plasma PK parameters (AUC(0-t), Cmax) of daprodustat

#### **Model Specification (Part 1)**

#### Part 1

 The exposure (AUC(0-t) and Cmax) of daprodustat will be assessed by using a mixed effect model as described below:

```
log<sub>e</sub> (PK parameter) = \beta_0 + \gamma_i + \tau_j + \pi_k + \alpha_l + \epsilon_{ijkl}

\beta_0: intercept

\gamma_i: random subject effect for ith subject, following N(0, \sigma_b^2)

\tau_j: tablet strength effect (j = 2 mg or 4 mg)

\pi_k: period effect (k = period 1 or period 2)

\alpha_l: group effect (l= group A or group B)

\epsilon_{ijkl}: random error for subject i, tablet strength j, period k, group I, following N(0, \sigma_w^2)
```

- The model parameters will be estimated using Restricted Maximum Likelihood with the Newton-Raphson algorithm.
- The Kenward-Roger degree of freedom approach will be used.
- Given the random effect for subject i, the random error is assumed to be independently distributed within the subject.
- The least square means for each tablet strength will be estimated based on the fitted model.
   The mean difference between tablet strengths (2mg 4mg) and its 90% CIs will be also estimated using the within-subject variance.
- The estimates of least square means for each tablet strength, the treatment difference between tablet strength and the 90% CIs will be exponentially back-transformed to obtain the estimates of geometric means of AUC(0-t) and Cmax for each tablet strength, the ratio of geometric means (2mg/4mg) and its 90% CIs, respectively.
- Within-subject variability (%CVw) for the PK parameters will be estimated using within-subject variance from the analysis model as follows:

%CVw (%) = 
$$[exp(\sigma_w^2) - 1]^{1/2} \times 100$$

AUC(0-inf) will be analyzed in the same manner.

#### Part 2

 To estimate the food effect on PK parameters (AUC(0-t) and Cmax) of daprodustat, the PK parameters will be analysed using a mixed effect model as described as below (almost the same as Part 1):

```
log<sub>e</sub> (PK parameter) = \beta_0 + \gamma_i + \tau_j + \pi_k + \alpha_l + \epsilon_{ijkl}

\beta_0: intercept

\gamma_i: random subject effect for ith subject

\tau_i: food effect (j = fed or fasted)
```

- $\pi_k$ : period effect (k = period 1 or period 2)  $\alpha_l$ : group effect (l= group C or group D)  $\epsilon_{ijkl}$ : random error for subject i, food effect i, period k, group l.
- The model restrictions will be the same as Part 1.
- The way of construction for the estimates of summary statistics will be the same as Part 1
  - Note that the ratio of geometric means (fed/fasted) and its 90% CIs for AUC(0-t) and Cmax will be estimated.
  - o AUC(0-inf) will be analyzed in the same manner.

#### **Model Checking & Diagnostics**

• In case there is a problem with model convergence, the arithmetic means for loge-transformed AUC(0-t) and Cmax and the treatment differences (2mg - 4mg in Part 1, fed - fasted in Part 2) within each subject will be calculated using only data from the subjects who have completed both 2mg and 4mg in Part 1, or both fed and fasted in Part 2. The mean treatment difference and paired-t test based 90% CIs for treatment difference in loge scale will be estimated. The results will be provided in an exponentially back-transformed scale.

#### **Model Results Presentation**

#### Part 1 and Part 2

- Results of Part 1 and Part 2 will be presented in the same manner, separately.
- The estimates of geometric means of PK parameters (AUC(0-t) and Cmax) will be presented
  for each tablet strength (Part 1) or for each food state (Part 2), respectively. The estimates of
  the geometric means ratio between tablet strengths (Part 1) or between fed and fasted state
  (Part 2) will be presented along with the associated 90% CIs and %CVw.
- For Part 1, the bioequivalence between daprodustat 2 mg tablet and 4 mg tablet will be evaluated as follows:
  - The bioequivalence is established when the 90% CI of the ratio for AUC(0-t) and Cmax between tablet strength (2 mg x 2 vs. 4 mg x 1) are within the range of 0.80 to 1.25.
  - Even if the 90% CI doesn't meet the above criteria, the bioequivalence is established when the point estimate of the ratio for AUC(0-t) and Cmax between tablet strength (2 mg x 2 vs. 4 mg x 1) are within the range of 0.90 to 1.11.
- AUC(0-inf) will also be provided in the model results presentation, but the evaluation of the bioequivalence will not be done based on AUC(0-inf).

## 8.1.6. Details of Planned Pharmacokinetic Displays

Summaries will be provided by Part (2mg tablet x 2 and 4mg tablet x 1 in Part 1, fed state and fasted state in Part 2), unless otherwise specified.

#### <u>Daprodustat Plasma Concentration-Time Data</u>

Daprodustat plasma concentrations at every scheduled time point will be summarized using n, mean, standard deviation, median, minimum, and maximum.

#### Derived Daprodustat Plasma Pharmacokinetic Parameters (non-transformed)

Daprodustat plasma pharmacokinetic parameters (AUC(0-t), AUC(0-inf), Cmax, Tmax, t1/2, %AUCex, CL/F, Vz/F, kel, and MRT) will be summarized using n, mean, 95% CI, standard deviation, median, minimum, and maximum.

#### Derived Daprodustat Plasma Pharmacokinetic Parameters (log-transformed)

For each pharmacokinetic parameters with a log-normal distribution (AUC(0-t), AUC(0-inf), Cmax, t1/2, %AUCex, CL/F, Vz/F, kel, and MRT), the log-transformed parameters will be summarized using n, geometric mean, 95% CI of geometric mean, standard deviation of log-transformed data and between subject coefficient of variation (%CVb).

### Analysis of Tablet Strength/Food Effect for AUC(0-t) and Cmax

The analysis results will be presented as described in Section 8.1.5.1 - *Model Results Presentation*. AUC(0-inf) will also be analysed and provided in a display.

# 9. REFERENCES

GlaxoSmithKline Document Number 2017N354137\_00 Study ID 207727. A single centre, single dose, open-label, randomised, 2-way crossover study in healthy Japanese male subjects to evaluate the bioequivalence of daprodustat tablets (2 mg tablet vs. 4 mg tablet) (Part 1) and the food effect on the pharmacokinetics of daprodustat (Part 2). Report Date 12-Mar-2018.

Japanese Society of Nephrology. Dietary recommendations for chronic kidney disease, 2014. Jpn J Nephrol. 2014;56(5):533-59.

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the PDMP and the data handling will be determined prior to DBR.

# 10.2. Appendix 2: Schedule of Activities

#### 10.2.1. Protocol Defined Schedule of Events

| | C | Intervention period (Period 1-2) | | | | | | | | | | | | | F-11 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Scree<br>ning <sup>1</sup> | Day | Day Day 1 | | | | | | | | | | | Day 2 | Follow-<br>up <sup>7</sup> | |
| | illig | -1 | Pre-dose | 0 h | 0.5 h | 1 h | 1.5 h | 2 h | 2.5 h | 3 h | 4 h | 6 h | 8 h | 12 h | 24 h | ир |
| Informed consent | Χ | | | | | | | | | | | | | | | |
| Demography/Medical history | Χ | | | | | | | | | | | | | | | |
| Height, Weight, Body mass index (BMI) | Χ | | | | | | | | | | | | | | | |
| Urine drug screen | Χ | | | | | | | | | | | | | | | |
| Serology test <sup>2</sup> | Χ | | | | | | | | | | | | | | | |
| Physical examination | Χ | Χ | Х | | | | | | | Χ | | | | | Χ | Χ |
| 12-lead ECG | Χ | | Х | | | | | | | Χ | | | | | Χ | Χ |
| Vital signs <sup>3</sup> | Χ | | Х | | | | | | | Х | | | | | Χ | Х |
| Clinical laboratory test <sup>4</sup> | Χ | Χ | | | | | | | | | | | | | Χ | Χ |
| Study intervention dosing <sup>5</sup> | | | | Χ | | | | | | | | | | | | |
| PK blood sampling | | | Х | | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | |
| AE <sup>6</sup> /Serious adverse events (SAE) <sup>6</sup> | <==== | ===== | | | ====== | ===== | ====== | ===== | | ====== | | ===== | | | ====== | =====> |
| Concomitant medication review | <==== | | | | | =====> | | | | | | | | | | |
| Admission to unit | | Χ | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | Χ | |
| Outpatient visit | Χ | | | | | | | | | | | | | | | Х |

- 1: Within 30 days prior to Day 1 of Period 1.
- 2: Serology tests for syphilis [Rapid plasma reagin (RPR) & Treponema pallidum (TP)], Human immunodeficiency virus (HIV) antigen/antibody, Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody and Human T-cell lymphotropic virus type 1 (HTLV-1) antibody.
- 3: Body temperature (axillary), systolic and diastolic blood pressure and pulse (supine).
- 4: Haematology, clinical chemistry and urinalysis.
- 5: Subjects will remain in a sitting or semi-supine position for approximately 4 hours if possible after dosing on Day 1. In Part 2, study subjects who are in fed state should take a standard meal as recommended for chronic kidney disease (CKD) by the Japanese Society of Nephrology in Japan [Jpn J Nephrol, 2014] in 20 minutes or less and the drug product should be administered 30 minutes after the end of the meal.
- 6: AEs and SAEs will be collected from the start of intervention until the follow-up visit at the time points specified. However, any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, or invasive tests) will be recorded from the time a subject consents to participate in the study.
- 7: 7(±1) days post-dose of Period 2.

# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 10.3.1. Study Phases

Assessments and events (e.g., study withdrawal) will be classified according to the time of occurrence relative to dosing start Date and Time by Period. The following definitions will be applicable to both Part 1 and Part 2.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Reference Day < Previous Day of Dosing Start Date in Period 1 |
| Period 1 | Previous Day of Dosing Start Date in Period 1 ≤ Reference Day < Previous Day of Dosing Start Date in Period 2 |
| Period 2 | Previous Day of Dosing Start Date in Period 2 ≤ Reference Day |

#### 10.3.1.1. Study Phases for Adverse Events

The study phases for AEs will be categorized into pre-treatment, period 1, and period 2 based on AE onset date and time.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | AE Onset Date and Time < Study First Dosing Start Date and Time |
| Period 1 | Study First Dosing Start Date and Time ≤ AE Onset Date and Time < Dosing Start Date and Time in Period 2 |
| Period 2 | Dosing Start Date and Time in Period 2 ≤ AE Onset Date and Time |
| Time since Study<br>First Dose (min) | If study phase of the event is pre-treatment, AE Onset Date and Time - Study First Dosing Start Date and Time otherwise AE Onset Date and Time - Study First Dosing Start Date and Time + 1 min |
| Time since Period<br>First Dose (min) | If study phase of the AE is pre-treatment, set to missing If study phase of the AE is period 1, AE Onset Date and Time – Dosing Start Date and Time in Period 1 + 1 min If study phase of the AE is period 2, AE Onset Date and Time – Dosing Start Date and Time in Period 2 + 1 min |
| Time since Last<br>Dose (min) | If study phase of the AE is pre-treatment, set to missing If AE Onset Date and Time ≥ Study Last Dosing Start Date and Time, AE Onset Date and Time – Study Last Dosing Start Date and Time+ 1 min |
| Duration (min) | AE Resolution Date and Time – AE Onset Date and Time + 1 min |
| Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be treatment emergent.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.3.1.2. Study Phases for Concomitant Medication

The study phases for concomitant medications represent the period of medication star. The study phases will be categorized into pre-treatment, period 1, and period 2 based on medication start date and time.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Start Date and Time < Study First Dosing Start Date and Time |
| Period 1 | Study First Dosing Start Date and Time ≤ Start Date and Time < Dosing Start Date and Time in Period 2 |
| Period 2 | Dosing Start Date and Time in Period 2 ≤ Start Date and Time |

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

## 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : N/A |
| HARP Compound | : N/A |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated. | |

### 10.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visit**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Office will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | No PK parameters derived by programmer are planned. : |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters in GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards: Standards for the Transfer and Reporting of PK Data using HARP |

## 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dosing Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dosing Date → Study Day = Ref Date First Dosing Date
- Ref Date ≥ First Dosing Date → Study Day = Ref Date (First Dosing Date) + 1

#### **Period Day**

- Calculated as the number of days from Dosing Date in Period 1 or Period 2.
  - If Study Phase of Ref Assessment or Event = Pre-Treatment or Missing
    - → Period Day = Missing
  - If Study Phase of Ref Assessment or Event = Period 1
    - → If Ref Date is on or after Dosing Date in Period 1, Period Day = Ref Date Dosing Date in Period 1 + 1 day
    - → If Ref Date is before Dosing Date in Period 1, Period Day = Ref Date Dosing Date in Period 1
  - If Study Phase of Ref Assessment or Event = Period 2
    - → If Ref Date is on or after Dosing Date in Period 2, Period Day = Ref Date Dosing Date in Period 2 + 1 day
    - → If Ref Date is before Dosing Date in Period 2, Period Day = Ref Date Dosing Date in Period 1

## 10.5.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - A date and month will be imputed as '30th June' as it will not be captured.
- Date of Informed Consent will be used as reference date of calculation.

## 10.5.3. Safety

#### **Laboratory Parameters**

#### **Imputation**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

o Example 1: 2 Significant Digits = '< x' becomes x - 0.01o Example 2: 1 Significant Digit = '> x' becomes x + 0.1o Example 3: 0 Significant Digits = '< x' becomes x - 1

 The default convention for reporting of clinical laboratory units will be the international system of units (SI units).

#### PCI

• For PCI listings of the absolute neutrophils and lymphocytes count, PCI cutoffs will be calculated by multiplying the percentages given for each subject by the absolute white blood count.

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study including the follow up visit.</li> <li>If subjects prematurely withdraw from the study, additional replacement participants may be recruited and assigned to the same treatment sequence.</li> </ul> |
| | <ul> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.6.2.1. Handling of Missing and Partial Dates and Times

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> </ul> |
| Adverse<br>Events | <ul> <li>The eCRF does not allow for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month will not be missing.</li> <li>The eCRF allows for the possibility of missing times to be recorded for AE start and end dates. Missing times will be imputed using the following convention: <ul> <li>If the missing time is a start time, a '00:00' will be used for the time.</li> <li>If the missing time is a stop time, a '23:59' will be used for the time.</li> </ul> </li> <li>The recorded missing time will be displayed in listings without imputed values.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The eCRF allows for the possibility of missing times to be recorded for concomitant medications start and end dates. Missing times will be imputed using the following convention:</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>If the missing time is a start time, a '00:00' will be used for the time.</li> </ul> |
| | <ul> <li>If the missing time is a stop time, a '23:59' will be used for the time.</li> </ul> |
| | The recorded partial date and missing time will be displayed in listings without imputed values. |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Haamataarit | Ratio of | | | 0.54 |
| Haematocrit | 1 | $\Delta$ from BL | ↓0.075 | |
| Haamaglahin | g/L | | | 180 |
| Haemoglobin | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Cell Count | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | μmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |
# 10.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 10.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Con | cern Range |
|--------------------------|-------|--------------|------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.8. Appendix 8: Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| AST | Aspartate transaminase |
| AUC(0-inf) | Area under the concentration-time curve from time zero (pre-dose) extrapolated |
| 7.00(0) | to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last time |
| , | of quantifiable concentration within a subject across all treatments |
| BL | Baseline |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CSR | Clinical Study Report |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| MRT | Mean Residence Time |
| NQ | Non-quantifiable |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RTF | Rich Text File |
| SAC | Statistical Analysis Complete |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| SOP | Standard Operation Procedure |
| t1/2 | Terminal half-life |
| Tmax | Time to maximum observed blood drug concentration |
| TFL | Tables, Figures & Listings |
| ULN | Upper Limit of Normal |
| WNL | WinNonlin |

# 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

## 10.9. Appendix 9: List of Data Displays

### 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------------------|----------------|
| Study Population | 1.1 to 1.9 | Not Applicable |
| Safety | 2.1 to 2.36 | Not Applicable |
| Pharmacokinetic | 3.1 to 3.8 3.1 to 3.10 | |
| Section | Listings | |
| ICH Listings | 1 to 75 | |

## 10.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | jure Table I | |
|-----------------|--------|--------------|-------|
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.9.3. Deliverables

| <b>Delivery Priority</b> | Description |
|--------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.9.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Subjec | ct Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Subject Disposition (Part 1) | ICH E3, FDAAA, EudraCT Only total column will appear | SAC |
| 1.2. | Safety | ES1A | Summary of Subject Disposition (Part 2) | ICH E3, FDAAA, EudraCT<br>Only total column will appear | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements Only total column will appear. Not provided separately by Part | SAC |
| 1.4. | Enrolled | NS1 | Summary of Number of Subject by Country and Site ID | EudraCT/Clinical Operations Only total column will appear. Not provided separately by Part | SAC |
| Protoc | ol Deviation | | | | |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations (Part 1) | ICH E3 Only total column will appear | SAC |
| 1.6. | Safety | DV1 | Summary of Important Protocol Deviations (Part 2) | ICH E3 Only total column will appear | SAC |
| Demo | graphic and Bas | seline Characteris | tics | | |
| 1.7. | Safety | DM3 | Summary of Demographic Characteristics (Part 1) | ICH E3, FDAAA, EudraCT Only total column will appear | SAC |
| 1.8. | Safety | DM3 | Summary of Demographic Characteristics (Part 2) | ICH E3, FDAAA, EudraCT<br>Only total column will appear | SAC |
| 1.9. | Enrolled | DM11 | Summary of Age Ranges | EudraCT/Clinical Operations Only total column will appear. Not provided separately by Part | SAC |

207727

# 10.9.5. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | • |
| 2.1. | Safety | AE1CP | Summary of All AE by SOC and PT (Part 1) | ICH E3<br>Include total column | SAC |
| 2.2. | Safety | AE1CP | Summary of All AE by SOC and PT (Part 2) | ICH E3<br>Include total column | SAC |
| 2.3. | Safety | AE5A | Summary of All AEs by Maximum Intensity by SOC and PT (Part 1) | ICH E3<br>Include total column | SAC |
| 2.4. | Safety | AE5A | Summary of All AEs by Maximum Intensity by SOC and PT (Part 2) | ICH E3<br>Include total column | SAC |
| 2.5. | Safety | AE1CP | Summary All Drug-Related AE by SOC and PT (Part 1) | ICH E3<br>Include total column | SAC |
| 2.6. | Safety | AE1CP | Summary All Drug-Related AE by SOC and PT (Part 2) | ICH E3<br>Include total column | SAC |
| 2.7. | Safety | AE5A | Summary of All Drug-Related AEs by Maximum Intensity by SOC and PT (Part 1) | ICH E3<br>Include total column | SAC |
| 2.8. | Safety | AE5A | Summary of All Drug-Related AEs by Maximum Intensity by SOC and PT (Part 2) | ICH E3<br>Include total column | SAC |
| Labora | tory: Chemistry | / | | | |
| 2.9. | Safety | LB1 | Summary of Chemistry Data (Part 1) | | SAC |
| 2.10. | Safety | LB1 | Summary of Chemistry Data (Part 2) | | SAC |
| 2.11. | Safety | LB1 | Summary of Chemistry Change from Baseline (Part 1) | ICH E3 Include baseline value | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | Safety | LB1 | Summary of Chemistry Change from Baseline (Part 2) | ICH E3 Include baseline value | SAC |
| 2.13. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline Relative to Normal Range (Part 1) | ICH E3 | SAC |
| 2.14. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline Relative to Normal Range (Part 2) | ICH E3 | SAC |
| Labora | tory: Haematol | ogy | | <u>'</u> | |
| 2.15. | Safety | LB1 | Summary of Haematology Data (Part 1) | | SAC |
| 2.16. | Safety | LB1 | Summary of Haematology Data (Part 2) | | SAC |
| 2.17. | Safety | LB1 | Summary of Haematology Change from Baseline (Part 1) | ICH E3 Include baseline value | SAC |
| 2.18. | Safety | LB1 | Summary of Haematology Change from Baseline (Part 2) | ICH E3 Include baseline value | SAC |
| 2.19. | Safety | LB4 | Summary of Haematology Data Shifts from Baseline Relative to Normal Range (Part 1) | ICH E3 | SAC |
| 2.20. | Safety | LB4 | Summary of Haematology Data Shifts from Baseline Relative to Normal Range (Part 2) | ICH E3 | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | • |
| 2.21. | Safety | LB1 | Summary of Urinalysis Data (Gravity and pH) (Part 1) | | SAC |
| 2.22. | Safety | LB1 | Summary of Urinalysis Data (Gravity and pH) (Part 2) | | SAC |
| 2.23. | Safety | LB1 | Summary of Urinalysis Change from Baseline (Gravity and pH) (Part 1) | ICH E3<br>Include baseline value | SAC |
| 2.24. | Safety | LB1 | Summary of Urinalysis Change from Baseline (Gravity and pH) (Part 2) | ICH E3<br>Include baseline value | SAC |

| Safety | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | ulation IDSL / Example Shell Title P | | Programming Notes | Deliverable [Priority] |
| 2.25. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) (Part 1) | | SAC |
| 2.26. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) (Part 2) | SAC | |
| ECG | | | | | |
| 2.27. | Safety | EG1 | Summary of ECG Findings (Part 1) | IDSL | SAC |
| 2.28. | Safety | EG1 | Summary of ECG Findings (Part 2) | IDSL | SAC |
| 2.29. | Safety | EG2 | Summary of ECG Values (Part 1) | IDSL | SAC |
| 2.30. | Safety | EG2 | Summary of ECG Values (Part 2) | IDSL | SAC |
| 2.31. | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 1) | IDSL<br>Include baseline value | SAC |
| 2.32. | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 2) | IDSL<br>Include baseline value | SAC |
| Vital S | igns | | | | |
| 2.33. | Safety | VS1 | Summary of Vital Signs (Part 1) | IDSL | SAC |
| 2.34. | Safety | VS1 | Summary of Vital Signs (Part 2) | IDSL | SAC |
| 2.35. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 1) | ICH E3 Include baseline value | SAC |
| 2.36. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 2) | ICH E3 Include baseline value | SAC |

207727

### 10.9.6. Pharmacokinetic Tables

| Pharma | acokinetic: Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>Priority |
| 3.1. | PK | PK01 | Summary of Daprodustat Plasma Concentration-Time Data (Part 1) | | SAC |
| 3.2. | PK | PK01 | Summary of Daprodustat Plasma Concentration-Time Data (Part 2) | | SAC |
| 3.3. | PK | PK03 | Summary of Derived Daprodustat Plasma Pharmacokinetic Parameters (non-transformed) (Part 1) | | SAC |
| 3.4. | PK | PK03 | Summary of Derived Daprodustat Plasma Pharmacokinetic Parameters (non-transformed) (Part 2) | | SAC |
| 3.5. | PK | PK05 | Summary of Derived Daprodustat Plasma Pharmacokinetic Parameters (log-transformed) (Part 1) | | SAC |
| 3.6. | PK | PK05 | Summary of Derived Daprodustat Plasma Pharmacokinetic Parameters (log-transformed) (Part 2) | | SAC |
| 3.7. | PK | PK_T1 | Analysis of Tablet Strength Effect for Cmax, AUC(0-t), and AUC(0-inf) (Part 1) | Example Shell in Appendix 10 | SAC |
| 3.8. | PK | PK_T1 | Analysis of Food Effect for Cmax, AUC(0-t), and AUC(0-inf) (Part 2) | Example Shell in Appendix 10 | SAC |

# 10.9.7. Pharmacokinetic Figures

| Pharma | acokinetic: Figi | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.1. | PK | PK16b | Individual Daprodustat Plasma Concentration-Time Plots by Subject (Part 1) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.2. | PK | PK16b | Individual Daprodustat Plasma Concentration-Time Plots by Subject (Part 2) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.3. | PK | PK16b | Individual Daprodustat Plasma Concentration-Time Plots by Tablet Strength (Part 1) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.4. | PK | PK16b | Individual Daprodustat Plasma Concentration-Time Plots by Food State (Part 2) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.5. | PK | PK17 | Mean (+SD) Daprodustat Plasma Concentration-Time Plots (Part 1) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.6. | PK | PK17 | Mean (+SD) Daprodustat Plasma Concentration-Time Plots (Part 2) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.7. | PK | PK18 | Median Daprodustat Plasma Concentration-Time Plots (Part 1) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.8. | PK | PK18 | Median Daprodustat Plasma Concentration-Time Plots (Part 2) | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.9. | PK | PK_F1 | Plot of Individual Daprodustat Plasma Cmax, AUC(0-t), and AUC(0-inf) by Tablet Strength (Part 1) | Example Shell in Appendix 10 | SAC |
| 3.10. | PK | PK_F1 | Plot of Individual Daprodustat Plasma Cmax, AUC(0-t), and AUC(0-inf) by Food State (Part 2) | Example Shell in Appendix 10 | SAC |

207727

# 10.9.8. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | | Programming Notes | Deliverable<br>[Priority] |
| Study | Population | | | | • |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines Not provided separately | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal (Part 1) | ICH E3 | SAC |
| 3. | Safety | ES3 | Listing of Reasons for Study Withdrawal (Part 2) | ICH E3 | SAC |
| 4. | Safety | SD3 | Listing of Reasons for Treatment Discontinuation (Part 1) | ICH E3 | SAC |
| 5. | Safety | SD3 | Listing of Reasons for Treatment Discontinuation (Part 2) | ICH E3 | SAC |
| 6. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 1) | IDSL | SAC |
| 7. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 2) | IDSL | SAC |
| Protoc | ol Deviations | | | | <u>.</u> |
| 8. | Safety | DV2A | Listing of Important Protocol Deviations (Part 1) | ICH E3 | SAC |
| 9. | Safety | DV2A | Listing of Important Protocol Deviations (Part 2) | ICH E3 | SAC |
| 10. | Safety | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part 1) | ICH E3 | SAC |
| 11. | Safety | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part 2) | ICH E3 | SAC |
| Popula | tions Analysed | 1 | | | |
| 12. | Safety | SP3A | Listing of Subjects Excluded from PK Population (Part 1) | ICH E3 | SAC |
| 13. | Safety | SP3A | Listing of Subjects Excluded from PK Population (Part 2) | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | seline Characteris | tics | | <u>.</u> |
| 14. | Safety | DM4 | Listing of Demographic Characteristics (Part 1) | ICH E3 | SAC |
| 15. | Safety | DM4 | Listing of Demographic Characteristics (Part 2) | ICH E3 | SAC |
| 16. | Safety | DM10 | Listing of Race (Part 1) | ICH E3 | SAC |
| 17. | Safety | DM10 | Listing of Race (Part 2) | ICH E3 | SAC |
| Prior a | nd Concomitar | t Medications | | • | · |
| 18. | Safety | MH3 | Listing of Medical Conditions (Part 1) | IDSL | SAC |
| 19. | Safety | MH3 | Listing of Medical Conditions (Part 2) | IDSL | SAC |
| 20. | Safety | CM5 | Listing of Concomitant Medications (Part 1) | IDSL | SAC |
| 21. | Safety | CM5 | Listing of Concomitant Medications (Part 2) | IDSL | SAC |
| Exposi | ure | | | | · |
| 22. | Safety | EX4 | Listing of Exposure Data (Part 1) | ICH E3 | SAC |
| 23. | Safety | EX4 | Listing of Exposure Data (Part 2) | ICH E3 | SAC |
| Meal | | | | | · |
| 24. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days (Part 2) | | SAC |
| Safety | | | | | <u>.</u> |
| Advers | se Events | | | | |
| 25. | Safety | AE9CP | Listing of All Adverse Events (Part 1) | ICH E3 | SAC |
| 26. | Safety | AE9CP | Listing of All Adverse Events (Part 2) | ICH E3 | SAC |
| 27. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 1) | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 28. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 2) | ICH E3 | SAC |
| 29. | Safety | AE2 | Listing of Relationship between System Organ Class and Verbatim Text | IDSL<br>Not provided separately | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 30. | Safety | AE9CPa | Listing of Serious Adverse Events (Part 1) | ICH E3 | SAC |
| 31. | Safety | AE9CPa | Listing of Serious Adverse Events (Part 2) | ICH E3 | SAC |
| 32. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Part 1) | ICH E3 | SAC |
| 33. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Part 2) | ICH E3 | SAC |
| 34. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 1) | ICH E3 | SAC |
| 35. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 2) | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 36. | Safety | МН3 | Listing of Medical Conditions for Participants with Liver Stopping Events (Part 1) | IDSL | SAC |
| 37. | Safety | МН3 | Listing of Medical Conditions for Participants with Liver Stopping Events (Part 2) | IDSL | SAC |
| 38. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events (Part 1) | IDSL | SAC |
| 39. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events (Part 2) | IDSL | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | · |
| 40. | Safety | LB6 | Listing of All Chemistry Data (Part 1) | | SAC |
| 41. | Safety | LB6 | Listing of All Chemistry Data (Part 2) | | SAC |
| 42. | Safety | LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | ICH E3 | SAC |
| 43. | Safety | LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | ICH E3 | SAC |
| 44. | Safety | LB6 | Listing of All Haematology Data (Part 1) | | SAC |
| 45. | Safety | LB6 | Listing of All Haematology Data (Part 2) | | SAC |
| 46. | Safety | LB6 | Listing of All Haematology Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | ICH E3 | SAC |
| 47. | Safety | LB6 | Listing of All Haematology Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | ICH E3 | SAC |
| 48. | Safety | LB6 | Listing of Chemistry Values of Potential Clinical Importance (Part 1) | | SAC |
| 49. | Safety | LB6 | Listing of Chemistry Values of Potential Clinical Importance (Part 2) | | SAC |
| 50. | Safety | LB6 | Listing of Haematology Values of Potential Clinical Importance (Part 1) | | SAC |
| 51. | Safety | LB6 | Listing of Haematology Values of Potential Clinical Importance (Part 2) | | SAC |
| 52. | Safety | LB6 | Listing of Urinalysis Data (gravity and pH) (Part 1) | | SAC |
| 53. | Safety | LB6 | Listing of Urinalysis Data (gravity and pH) (Part 2) | | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Shell | | sulation Title D | | Deliverable<br>[Priority] |
| 54. | Safety | LB14 | Listing of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) (Part 1) | ICH E3 | SAC |
| 55. | Safety | LB14 | Listing of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) (Part 2) | ICH E3 | SAC |
| ECG | | | | | · |
| 56. | Safety | EG4 | Listing of All ECG Values (Part 1) | | SAC |
| 57. | Safety | EG4 | Listing of All ECG Values (Part 2) | | SAC |
| 58. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part 1) | IDSL | SAC |
| 59. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part 2) | IDSL | SAC |
| 60. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance (Part 1) | IDSL | SAC |
| 61. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance (Part 2) | IDSL | SAC |
| 62. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding (Part 1) | IDSL | SAC |
| 63. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding (Part 2) | IDSL | SAC |
| 64. | Safety | EG6 | Listing of Abnormal ECG Findings (Part 1) | IDSL | SAC |
| 65. | Safety | EG6 | Listing of Abnormal ECG Findings (Part 2) | IDSL | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | ation IDSL / Example Shell Title | | Programming Notes | Deliverable [Priority] |
| Vital Si | gns | | | | |
| 66. | Safety | VS5 | Listing of All Vital Signs Data (Part 1) | IDSL | SAC |
| 67. | Safety | VS5 | Listing of All Vital Signs Data (Part 2) | IDSL | SAC |
| 68. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | IDSL | SAC |
| 69. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | IDSL | SAC |
| 70. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance (Part 1) | IDSL | SAC |
| 71. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance (Part 2) | IDSL | SAC |
| PK | | | | | |
| 72. | PK | PK08 | Listing of Daprodustat Plasma Pharmacokinetic Concentration-<br>Time Data (Part 1) | IDSL | SAC |
| 73. | PK | PK08 | Listing of Daprodustat Plasma Pharmacokinetic Concentration-<br>Time Data (Part 2) | IDSL | SAC |
| 74. | PK | PK14 | Listing of Derived Daprodustat Plasma Pharmacokinetic Parameters (Part 1) | IDSL All PK parameters in Section 8.1.1.2 will be provided in a listing | SAC |
| 75. | PK | PK14 | Listing of Derived Daprodustat Plasma Pharmacokinetic Parameters (Part 2) | IDSL All PK parameters in Section 8.1.1.2 will be provided in a listing | SAC |

207727

# 10.10. Appendix 10: Example Mock Shells for Data Displays

Example: PK T1 Page 1 of n

Protocol: 207727 Population: PK

| | | | | Adjusted | Ratio | | |
|---|---|---|---|---|---|---|---|
| Parameter | Treatment | N | n | Geom Mean | (trt2/trt1) | 90% CI | %CVw[1] |
| Cmax (unit) | trt1 | XX | XX | XX.XXX | X.XXX | (x.xxx, x.xxx) | X.XXX |
| | trt2 | XX | XX | XX.XXX | | | |
| AUC(0-t) (unit) | trt1 | XX | XX | XX.XXX | X.XXX | (x.xxx, x.xxx) | X.XXX |
| | trt2 | XX | XX | XX.XXX | | | |
| AUC(0-inf) (unit) | trt1 | XX | XX | XX.XXX | X.XXX | (x.xxx, x.xxx) | X.XXX |
| | trt2 | XX | XX | XX.XXX | | | |

<sup>[1]</sup> Within-subject variability of each PK parameter

Programming notes: For Part1, trt1 = "4mg x 1" and trt2 = "2mg x 2". For Part2, trt1 = "fasted" and trt2 = "fed".

207727

Example: PK\_F1 Page 1 of n

Protocol: 207727
Population: PK

Table X

Plot of Individual Daprodustat Plasma Cmax, AUC(0-t), AUC(0-inf) by [Tablet Strength Effect/Food Effect] (Part [1 or 2])



Note: Geometric mean and 95% CI

Programming notes: For Part1, trt1 = "4mg x 1" and trt2 = "2mg x 2". For Part2, trt1 = "fasted" and trt2 = "fed".

Programming notes: AUC(0-inf) will also be presented.

Programming notes: Figures will be presented in left (Cmax), center (AUC(0-t), and right (AUC(0-inf).